CLINICAL TRIAL: NCT01873781
Title: A Pilot Study Simulating Multifocal Intraocular Lenses in Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, assoc. Prof. Dr.med.univ., Medical University of Vienna
Other Study IDs: OPTH-200912
Record Dates: First submitted 2013-01-31; First posted 2013-06-10 (Estimated); Last update posted 2013-08-29 (Estimated); Status verified 2013-08

CONDITIONS: Lenses, Intraocular; Contrast Sensitivity; Visual Acuity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 30 healthy male and female subjects: 30 healthy male and female subjects aged 18-35
  Interventions: Drug: Cyclopentolatehydrochloride

INTERVENTIONS:
Drug: Cyclopentolatehydrochloride — Cyclopentolatehydrochloride 0.5% (Thilo, Alcon, Vienna), dose: 1 drop for study eye

SUMMARY:
Age related cataracts are responsible for about 51 percent of blindness worldwide and according to the WHO affect about 20 million people, according to the WH . As cataract surgery is firstline treatment in the western world, there is a constant attempt to improve artificial intraocular lenes (IOL).

As for this study, the investigators seek to compare four different IOL designs in in a psychophysiological setting, allowing to assess the impact of these IOLs on vision and psychological processing of visual information.

As these IOLs also have downsides, such as reduced light intensity or image alterations, the subjective preference and overall impression shall be investigated. The healthy subjects look through a stable spectacle frame mounted onto a table, which enables the investigator to insert the different IOLs. This would allow subjective testing of IOLs before surgery.

ELIGIBILITY:
Inclusion Criteria:

Men and women aged between 18 and 35 years

* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, between -1 and +1 diopters

Exclusion Criteria:

* > 0,5 diopters of cylinder
* Abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: young healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Eearly Treatment Diabetic Retinopathy Study (ETDRS) visual acuity score | 1 study day
  To investigate the psychophysiological impact of different optical setups on visual acuity at far, intermediate and near distance.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria